CLINICAL TRIAL: NCT07397923
Title: Evaluation of the Safety and Efficacy of the Digital Therapeutic Device Zenicom for Improving Aphasia in Patients With Subacute Stroke and Aphasia (AQ ≥25), a Multicenter, Single-blind, Prospective, Randomized Exploratory Clinical Trial
Brief Title: Exploratory Evaluation of the Digital Therapeutic Device Zenicom for Subacute Stroke Aphasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Konkuk University Hospital (Other); Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Kee Chang, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-2506-978-003
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aphasia; Stroke
Keywords: digital therapeutics; aphasia treatment; subacute stroke; korean language
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: A Multi-center randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: Conventional Speech Therapy + Digital Speech Therapy (Experimental): Performs conventional speech therapy for 30 minutes daily + additional digital speech therapy program during the 2-week treatment period.
  Interventions: Device: Zenicog; Other: Conventional Speech Therapy
- Control Group: Conventional Speech Therapy (Active Comparator): Performs only conventional speech therapy for 30 minutes daily during the 2-week treatment period.
  Interventions: Other: Conventional Speech Therapy

INTERVENTIONS:
Device: Zenicog — This medical device is a Software as a Medical Device (SaMD) consisting of a patient application and a patient management web portal for medical staff. It is designed to provide personalized digital therapeutic content to patients with aphasia for the alleviation and improvement of language function symptoms.
  The therapeutic mechanism of this device is speech therapy delivered through a personalized content program, intended to improve the language function of aphasia patients. The device's treatment program alleviates and improves language function based on Stimulation-Facilitation Treatment and Functional Communication techniques, which are aphasia speech therapy methods recommended by the Korean Clinical Practice Guidelines for Stroke Rehabilitation (Brain & Neurorehabilitation).
  The training recommendation model applied to this device provides personalized training content based on the subject's performance characteristics and proficiency level. The analyzed performance character
  Arms: Experimental Group: Conventional Speech Therapy + Digital Speech Therapy
Other: Conventional Speech Therapy — Conventional speech therapy is provided for 30 minutes daily in face-to-face by a Speech-Language-Pathologist

SUMMARY:
Clinical Trial Title A Multicenter, Single-Blind, Prospective, Randomized, Exploratory Clinical Trial to Evaluate the Safety and Efficacy of the Digital Therapeutic Device 'Zenicom' for Improving Aphasia in Patients with Subacute Stroke

Clinical Trial Objectives To evaluate the efficacy of the digital therapeutic device Zenicom.

To evaluate the safety of the digital therapeutic device Zenicom.

Clinical Trial Period 6 months from the date of clinical trial plan approval by the Ministry of Food and Drug Safety (MFDS).

Target Condition Patients with aphasia resulting from stroke lesions.

Target Sample Size Total of 20 subjects (10 in the experimental group and 10 in the control group).

Investigational Medical Device Zenicom

Clinical Trial Methodology

1. Device Information

   A) Experimental Device: Digital Speech Therapy Application

   Group: Performs conventional speech therapy for 30 minutes daily + additional digital speech therapy program during the 2-week treatment period.

   B) Control Device: Conventional Speech Therapy

   Group: Performs only conventional speech therapy for 30 minutes daily during the 2-week treatment period.
2. Treatment Duration:

   Total 2 weeks (10 working days; total usage of 600 minutes or more).
3. Visits:

Total of 3 visits including outpatient and therapy room visits.

Visit 1 (T-1): Screening

Visit 2 (T0): Baseline and Treatment initiation

Visit 3 (T1): Post-treatment assessment

Inclusion and Exclusion Criteria

1. Inclusion Criteria Patients who satisfy all of the following criteria:

   Adults aged 19 years or older.

   Patients confirmed by a specialist to have aphasia caused by a stroke lesion.

   Patients with first-ever subacute stroke (within 3 months of onset) diagnosed via radiological examination (CT, MRI).

   Patients diagnosed with aphasia based on the Speech Assessment (PK-WAB-R).

   Patients whose native language is Korean.

   Patients capable of voluntarily consenting to the study.
2. Exclusion Criteria Patients meeting any of the following criteria will be excluded:

Progressive or hemodynamically unstable stroke.

Patients with other neurological diseases suspected to affect language ability.

Co-morbid major psychiatric disorders requiring continuous medication (e.g., Major Depressive Disorder, Schizophrenia, Bipolar Disorder, Dementia).

Co-morbid major neurogenic diseases other than stroke.

Confirmed history of degenerative neuropathy.

Current or past substance or alcohol use disorder.

Visual impairment (Low vision severity: visual acuity of 0.1-0.3 or lower).

Intellectual disability.

Illiteracy (unable to read and consent).

Patients deemed inappropriate for participation for other reasons.

Refusal to participate in the study.

Suspension and Dropout Criteria

1. Suspension Criteria

   If circumstances observed during the trial make it judged unreasonable to continue the study.

   Occurrence of Serious Adverse Events (SAE).
2. Dropout Criteria

The subject requests to stop participation or withdraws consent during the trial.

The investigator determines that the subject cannot continue the trial due to adverse events (e.g., headache, eye fatigue, nausea, dizziness, etc.).

The subject arbitrarily takes medication expected to affect the comparative evaluation of the investigational device during the trial.

The dosage of medication that may affect the comparative evaluation of the investigational device is changed during the trial.

Discovery of major protocol violations, such as violation of inclusion/exclusion criteria.

The subject fails to attend scheduled visits and cannot be contacted.

The subject fails to perform the digital speech therapy program for a total of 600 minutes or more.

The investigator determines that the trial should be stopped for other reasons.

Endpoints (Outcome Measures)

1. Primary Efficacy Endpoint

   Change in PK-WAB-R scores between T0 and T1 between groups.
2. Secondary Efficacy Endpoints

Change in K-BNT scores between T0 and T1 between groups.

Change in K-SAQOL-12 scores between T0 and T1 between groups.

Statistical Analysis Methods To evaluate the change in PK-WAB-R between T0 and T1 between groups, an independent two-sample test will be used. Depending on the distribution of the change, a parametric method (Student's t-test) or a non-parametric method (Mann-Whitney U test) will be selected and applied.

To evaluate the changes in K-BNT and K-SAQOL-12 between T0 and T1 between groups, an independent two-sample test will be used. Depending on the distribution of the change, a parametric method (Student's t-test) or a non-parametric method (Mann-Whitney U test) will be selected and applied.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 years or older.
* Confirmed by a specialist to have aphasia caused by a stroke lesion.
* First-ever subacute stroke (within 3 months of onset) diagnosed via radiological examination (CT, MRI).
* Diagnosed with aphasia based on the Speech Assessment (PK-WAB-R).
* Whose native language is Korean.

Exclusion Criteria:

* Have progressive or hemodynamically unstable stroke.
* Having other neurological diseases suspected to affect language ability.
* Co-morbid major psychiatric disorders requiring continuous medication (e.g., Major Depressive Disorder, Schizophrenia, Bipolar Disorder, Dementia).
* Co-morbid major neurogenic diseases other than stroke.
* Confirmed history of degenerative neuropathy.
* Current or past substance or alcohol use disorder.
* Visual impairment (Low vision severity: visual acuity of 0.1-0.3 or lower).
* Intellectual disability.
* Illiteracy (unable to read and consent).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
PK-WAB AQ(Korean Version of PK-WAB-R AQ) | T-1: Screening T0: Baseline T1: EOT(end of treatment: 2week after)
  The Aphasia Quotient (AQ) is a weighted composite score derived from the Western Aphasia Battery (WAB) (or its Korean adaptation, PK-WAB-R). It serves as a primary quantitative index of the severity of spoken language deficits in patients with aphasia.

SECONDARY OUTCOMES:
K-BNT (Korean version of Boston Naming Test) | T-1: Screening T0: Baseline T1: EOT(end of treatment: 2week after)
  A standardized neuropsychological assessment tool designed to evaluate confrontation naming ability (lexical retrieval) in individuals with cognitive impairments. It is the linguistically and culturally adapted version of the widely used Boston Naming Test (BNT).
K-SAQoL-12 (Korean version of Stroke and Aphasia Quality of Life Scale-12) | T-1: Screening T0: Baseline T1: EOT(end of treatment: 2week after)
  K-SAQoL-12 is the shortened, validated Korean version of the Stroke and Aphasia Quality of Life Scale-39 (SAQoL-39). It is a patient-reported outcome measure (PROM) designed to assess Health-Related Quality of Life (HRQoL) specifically in stroke survivors with aphasia.
Adverse Event | T1: EOT(end of treatment: 2week after)
  Any adverse event occurred during intervention

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided